CLINICAL TRIAL: NCT02592278
Title: Prevention of Dental Caries Lesions With Fluoride Varnish in Erupting First Permanent Molars
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad Iberoamericana (Other)
Collaborators: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 04-2015
Record Dates: First submitted 2015-10-28; First posted 2015-10-30 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Dental Caries
Keywords: Dental Caries; Fluoride Varnish; Preschool child; Prevention
MeSH Terms: conditions — Dental Caries | interventions — sodium fluoride topical preparation; Sodium Fluoride; Control Groups; hydrated silica gel-based toothpaste

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fluoride Varnish each 6 months (Experimental): Fluoride Varnish application every 6 months.
  Interventions: Drug: Fluoride Varnish
- Fluoride Varnish each 3 months (Experimental): Fluoride Varnish application every 3 months.
  Interventions: Drug: Fluoride Varnish
- Fluoride tooth paste (Active Comparator): Control group. Twice a day brush with fluoride toothpaste.
  Interventions: Drug: Control Group

INTERVENTIONS:
Drug: Fluoride Varnish — Application of fluoride varnish every 3 and 6 months.
  Other Names: Duraphat (Colgate)
  Arms: Fluoride Varnish each 3 months; Fluoride Varnish each 6 months
Drug: Control Group — Twice a day brush with fluoride toothpaste.
  Other Names: Colgate Total Toothpaste
  Arms: Fluoride tooth paste

SUMMARY:
The aim of this study is to determine the effectiveness of fluoride varnishes in the prevention of dental caries lesions in erupting permanent first molars, in high-risk patients. Using as reference ICDAS criteria, when the success means that the surface maintain an ICDAS value 0 and failure that has change in ICDAS value 0 to 1.

Sample: The sample comprise 180 patients between 6-7 years old with high-risk of dental caries.

Study design: It proposed an experimental design randomized into 3 groups according to the frequency of topical fluoride application.(Group A: every 6 month; Group B: every 3 month; Group C: positive control).

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent from parents.
* Child assent
* High risk of dental caries
* At least one sound first permanent molar (ICDAS=0)

Exclusion Criteria:

* Bad behaviour
* Any systemic condition, disability

Ages: 6 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2015-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Number of first permanent molars with caries Lesion (taking into account ICDAS criteria) | One year
  We are going to measure changed to decay surfaces in first permanent molars = ICDAS > 0 in a year.

CONTACTS AND LOCATIONS:
Overall Officials: Ninoska Abreu, Principal Investigator — Universidad Iberoamericana